CLINICAL TRIAL: NCT03100812
Title: Asian American Partnerships in Research and Empowerment (AsPIRE)
Acronym: AsPIRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 07-1131
Record Dates: First submitted 2017-03-29; First posted 2017-04-04 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Hypertensive Heart Disease; Hypertension
Keywords: Hypertensive; Hypertension; Filipino
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental)
  Interventions: Behavioral: More intensive CHW Intervention
- Group B (Experimental)
  Interventions: Behavioral: Less Intensive CHW Intervention

INTERVENTIONS:
Behavioral: More intensive CHW Intervention — Group A participants will attend 4 monthly 90 minute group health education sessions that provide the tools and strategies to promote heart health to Filipino American individuals, families, and communities on high blood pressure and CVD. The CHWs will lead these sessions utilizing NHLBI's Healthy Heart Healthy Family, A CHW's Manual for the Filipino Community. Each of the group health education sessions will discuss different content related to CVD, hypertension, and other CVD risk factors. The first session focuses on assessing heart disease risk and recognition of heart attack signs. The second session focuses on physical activity and weight management and blood pressure control. The third session addresses control of cholesterol, and diabetes. The final 4th session teaches participants about nutrition and living smoke free.
  Arms: Group A
Behavioral: Less Intensive CHW Intervention — Individuals randomized to the less intensive CHW intervention will have the baseline, 4 month, and 8 month interviews and blood pressure measurements will be collected in those succeeding time points. Participants will also receive a 30 minute one on one session from the CHW and a referral to a physician if needed.
  Arms: Group B

SUMMARY:
The proposed intervention is part of a multi-year year grant awarded to the NYU Center for the Study of Asian American Health by to the National Institutes of Health/National Center for Minority Health and Health Disparities (NIH/NCMHD). The funding mechanism is specifically the NCMHD Community-Based Participatory Research (CBPR) Initiative in Reducing and Eliminating Health Disparities: Intervention Research Phase (R24).

The objective of this study is to implement and assess the efficacy of a Community Health worker (CHW) intervention to improve hypertension management and access to care among Filipino Americans living in New York and New Jersey. It is believed that when compared to individuals receiving the less intensive CHW intervention, Filipino Americans receiving the more intensive CHW intervention will:

H1: Exhibit greater compliance with appointment keeping. H2: Exhibit greater compliance with medication taking H3: Show greater reductions in mean systolic and mean diastolic blood pressure. H4: Be more likely to exhibit controlled blood pressure

DETAILED DESCRIPTION:
Filipino Americans exhibit high rates of hypertension and are therefore at high risk for cardiovascular disease and stroke. However, few interventions have been developed and implemented for this population to address these concerns. A CHW intervention, developed with community input to ensure its cultural and linguistic appropriateness, has the potential to prevent cardiovascular disease and stroke by helping Filipino Americans control their blood pressure. This study has the overall goal of improving health access and cardiovascular health status, particularly hypertension, in the Filipino American community living in New York City and New Jersey through the use of Community Health Workers (CHW).

ELIGIBILITY:
Inclusion Criteria:

* The population of interest is Filipino American men and women residing in New York City. An individual is eligible for the CHW intervention if he/she is

  1. of Filipino descent,
  2. an English or Tagalog-speaker
  3. a resident of New York City.
  4. identified as hypertensive based on
* The average of the 2nd and 3rd readings from both arms (right arm) with at least 1 high systolic BP (>140mmHg) or 1 high diastolic BP reading (>90mmHg) for nondiabetics, or 1 high systolic BP (>130mmHg) or 1 high diastolic BP reading (>80mmHg) for diabetics at point of screening for this study.
* Or if participant reports to be taking antihypertensive medication. Therefore this study will include individuals with untreated hypertension (not taking antihypertensive medication), uncontrolled hypertension (i.e. elevated blood pressure despite taking antihypertensive medication), and controlled hypertension (i.e. taking antihypertensive medication but BP is under control). Individuals presenting with untreated high blood pressure will be referred to a physician to confirm diagnosis of hypertension.

An individual is ineligible for enrollment in the CHW intervention if he/she

1. is on renal dialysis since their treatment is beyond the scope of this CHW intervention
2. has an acute or terminal illness or serious mental illness that deems an individual ineligible for study participation
3. is participating in another hypertension or CVD study
4. has had a history of a heart attack, stroke, or congestive heart failure, since their treatment is beyond the scope of this CHW intervention
5. has a blood pressure average below 140/90 for non-diabetics and not taking antihypertensive medication, and an average of 130/80 for diabetics not taking antihypertensive medication.
6. is below 25 or over 75 years of age
7. lives outside of NYC

Exclusion Criteria:

* An individual is ineligible for enrollment in the CHW intervention if he/she

  1. is on renal dialysis since their treatment is beyond the scope of this CHW intervention
  2. has an acute or terminal illness or serious mental illness that deems an individual ineligible for study participation
  3. is participating in another hypertension or CVD study
  4. has had a history of a heart attack, stroke, or congestive heart failure, since their treatment is beyond the scope of this CHW intervention
  5. has a blood pressure average below 140/90 for non-diabetics and not taking antihypertensive medication, and an average of 130/80 for diabetics not taking antihypertensive medication.
  6. is below 25 or over 75 years of age
  7. lives outside of NYC
* An individual is ineligible for enrollment in the CHW intervention if he/she

  1. is on renal dialysis since their treatment is beyond the scope of this CHW intervention
  2. has an acute or terminal illness or serious mental illness that deems an individual ineligible for study participation
  3. is participating in another hypertension or CVD study
  4. has had a history of a heart attack, stroke, or congestive heart failure, since their treatment is beyond the scope of this CHW intervention
  5. has a blood pressure average below 140/90 for non-diabetics and not taking antihypertensive medication, and an average of 130/80 for diabetics not taking antihypertensive medication.
  6. is below 25 or over 75 years of age
  7. lives outside of NYC
* An individual is ineligible for enrollment in the CHW intervention if he/she

  1. is on renal dialysis since their treatment is beyond the scope of this CHW intervention
  2. has an acute or terminal illness or serious mental illness that deems an individual ineligible for study participation
  3. is participating in another hypertension or CVD study
  4. has had a history of a heart attack, stroke, or congestive heart failure, since their treatment is beyond the scope of this CHW intervention
  5. has a blood pressure average below 140/90 for non-diabetics and not taking antihypertensive medication, and an average of 130/80 for diabetics not taking antihypertensive medication.
  6. is below 25 or over 75 years of age
  7. lives outside of NYC

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1000 (Actual)
Dates: Start 2010-09-23 (Actual); Primary Completion 2016-05-03 (Actual); Study Completion 2016-05-03 (Actual)

PRIMARY OUTCOMES:
Medication Adherance measured using the Hill-Bone Compliance to High Blood Pressure Therapy Scale | 12 Months
  This scale is comprised of 14 items in three subscales; one subscale pertains to adherence to medication taking. Three blood pressure readings will be taken; the second and third will be averaged.
Measures of Intensity and Fidelity of Community Health Worker Intervention | 12 Months
  Attendance at group sessions and individual home visits will be recorded to determine intervention dosage.

CONTACTS AND LOCATIONS:
Overall Officials: Chau Trinh, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

REFERENCES:
- [Derived] Wyatt LC, Katigbak C, Riley L, Zanowiak JM, Ursua R, Kwon SC, Trinh-Shevrin C, Islam NS. Promoting Physical Activity Among Immigrant Asian Americans: Results from Four Community Health Worker Studies. J Immigr Minor Health. 2023 Apr;25(2):291-305. doi: 10.1007/s10903-022-01411-y. Epub 2022 Oct 23. PMID 36273386